CLINICAL TRIAL: NCT06873386
Title: Effectiveness of Ultrasound-guided Percutaneous Electrical Stimulation of the Inferior and Superior Gluteal Nerves as Treatment for Gluteus Maximus and Medius Muscle Dysfunction After an Episode of Low Back Pain: Randomized Clinical Trial
Brief Title: Ultrasound-guided Percutaneous Electrical Stimulation for Gluteus Muscle Dysfunction After Low Back Pain Episode
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marc Badia (Other)
Responsible Party: Sponsor-Investigator, Marc Badia, physiotherapist, Universidad de Zaragoza
Organization: Universidad de Zaragoza (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.I. PI24/578
Record Dates: First submitted 2025-03-01; First posted 2025-03-12 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain; Functional Motor Disorder
Keywords: Low back pain; Muscle dysfunction; Neuromodulation; Nercutaneous ultrasound-guided neuromodulation; Neuromuscular activation; gluteal dysfunction after low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The principal investigator, who carries out the intervention, is not masked. The participants and the researchers in charge of analysing the outcome variables are masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valera & Minaya protocol (Active Comparator): US-guided PNM with the conventional frequency of the Valera Minaya protocol, with localised location on the peripheral nerve. Stimulation of the upper gluteal nerve and lower gluteal nerve will be performed, with 10 stimulations, with 10 seconds of stimulation and 10 seconds of rest, at a frequency of 10 Hz, with a pulse amplitude of 250 μs, and of maximum intensity tolerable by the patient that causes an exacerbated muscle contraction.
  Interventions: Device: Valera & Minaya protocol
- High-frequency PNM (Experimental): High-frequency US-guided PNM with localised peripheral nerve location. Ten 10-second stimulations of the upper gluteal nerve and lower gluteal nerve will be performed, with frequency sweeps of 20Hz -100Hz with a pulse amplitude of 250 μs, and of maximum intensity tolerable by the patient that causes an exacerbated muscle contraction, with 10 seconds of rest between each stimulation.
  Interventions: Device: High-frequency US-guided PNM

INTERVENTIONS:
Device: Valera & Minaya protocol — Valera & Minaya protocol:
  US-guided PNM with the conventional frequency of the Valera Minaya protocol, with localised location on the peripheral nerve. Stimulation of the upper gluteal nerve and lower gluteal nerve will be performed, with 10 stimulations, with 10 seconds of stimulation and 10 seconds of rest, at a frequency of 10 Hz, with a pulse amplitude of 250 μs, and of maximum intensity tolerable by the patient that causes an exacerbated muscle contraction.
  The specific device used will be an electric needle stimulator, AS Super 4 Digital, Schwa-medico Holistic Health, Ehringshausen, Germany.
  Other Names: convenctional frequency
  Arms: Valera & Minaya protocol
Device: High-frequency US-guided PNM — High-frequency US-guided PNM with localised peripheral nerve location. Ten 10-second stimulations of the upper gluteal nerve and lower gluteal nerve will be performed, with frequency sweeps of 20Hz -100Hz with a pulse amplitude of 250 μs, and of maximum intensity tolerable by the patient that causes an exacerbated muscle contraction, with 10 seconds of rest between each stimulation.
  The specific device used will be an electric needle stimulator, AS Super 4 Digital, Schwa-medico Holistic Health, Ehringshausen, Germany.
  Arms: High-frequency PNM

SUMMARY:
Percutaneous ultrasound-guided neuromodulation (US-guided PNM) is the electrical stimulation of a peripheral nerve at some point along its pathway or at a muscular motor point under the guidance of an ultrasound probe with a therapeutic objective.

The application of electrical current to a peripheral motor nerve is associated with a motor response that results in an uncontrolled, anarchic and exaggerated response of the musculature, which is normalized after the application of the electrical current.

In 2016, the authors of the book Invasive Physiotherapy, Fermín Valera and Francisco Minaya, developed by themselves based on the fundamentals of segmental dry needling and neurofunctional acupuncture created by Dr. Alejandro Elorriaga. The authors defined that the application parameters to achieve the best result to the electrical stimulus are controversial, due to the high variability in the literature, but knowing that the most important parameter is the frequency, where studies are observed in which they have used from 2 to 100Hz looking for the motor response.

The parameters of the protocol created are: frequency of 10Hz, pulse width of 250us, with a motor or sensory response, performing 8 stimulations of 8 seconds duration, with 8 seconds of rest, with the aim of improving neuromuscular function, muscle recruitment patterns and motor control.

Although the scientific basis of the authors were 3 articles, none of which were aimed at improving muscle function, but were for neuropathic pain, chronic pain, and treatment of overactive bladder, the basis of clinical observation is correct and many studies currently using their protocol show improvements at the functional level.

In a review of neuromodulation and muscle function, studies that carry out percutaneous stimulation use frequencies of 2Hz to 10Hz, using the protocol of Garrido F. V., Muñoz F. M. , which, as stated above, was not specifically designed to improve muscle function, while the studies that carry out transcutaneous stimulation use much higher frequencies, from 20Hz to 100Hz, all obtaining positive results.

For this reason, and the great difference between the frequencies, the need to carry out specific research on the benefits that percutaneous stimulation with a frequency range of 20-100 HZ.

The hypotheses of this study are,US-guided PNM, with frequency sweeps of 20Hz -100Hz increases static and dynamic strength, more relevantly than current 10Hz protocols.

DETAILED DESCRIPTION:
A randomised, double-blind, controlled clinical trial will be conducted in two parallel groups. Intervention group 1 will receive stimulation at 10Hz and intervention group 2 will receive stimulation with frequency sweeps of 20Hz-100Hz.

A period of pre-intervention baseline strength data collection is included to record gluteus maximus and gluteus minimus inhibition.

A single treatment intervention will be performed in the first week, with pre- and post-intervention assessment. Follow-up will last 4 weeks, with pre-intervention, post-intervention, 15 and 30 days post-intervention assessments.

This study follows the recommendations of the Consolidated Standards of Reporting Trials (CONSORT) statement for pragmatic clinical trials.

The objectives of this study are:

Primary objective:

To determine whether US-guided PNM with frequency sweeps of 20Hz-100Hz in inhibited musculature shows a greater response in dynamometrically measured static and dynamic force parameters than 10Hz stimuli.

Secondary objectives:

To analyse the duration of improvement in functional parameters. To analyse whether the patient tolerates the treatment better with stimuli with frequency sweeps of 20Hz-100Hz, than only with 10Hz stimuli.

Participants Users of both sexes of the Fiostec Funcional physiotherapy clinic in Sabadell, who have visited the clinic for an episode of low back pain in the last 2 years and who have also given their consent for the clinic to contact them for information purposes and who meet the inclusion criteria of the study, will be asked to participate.

Sample size To calculate the sample size, the minimum detectable change (MCD) in the dynamometric strength assessment was first calculated. For this purpose, data from a previous study were used, in which a standard error of measurement of 0.12 and an intraclass correlation coefficient of 0.91 were reported. With these data, a DCM of 0.33 points is obtained. Knowing the CMD, and adopting a conservative measure, it is decided to set the minimum clinically significant change (MCID) value at 1.30 points. This value is considerably higher than the CMD and corresponds to 10% of the mean strength (12.96) obtained in the previous study (https://pubmed.ncbi.nlm.nih.gov/35799746/). Using this MCID of 1.30 points, a standard deviation of 0.93, a significance level of 0.05 and a statistical power of 0.9, gives a required sample size of 24 participants to be included in this study.

Randomisation Subjects meeting the inclusion criteria will be randomly assigned to groups. The computer programme www.randomizer.org will be used.

Sources of information The personal data to be collected are: telephone number, name, age, type of work (static/dynamic), sex, number of episodes of low back pain, chronology of episodes of low back pain, laterality of lumbar involvement if any, sports practice or training. These data will be provided by the patient himself/herself on the first day he/she comes to the clinic.

The variables to be collected are: strength of the gluteus maximus and medius muscles in static and dynamic form with a dynamometer, surface electromyography. These variables will be recorded by the principal investigator, before and just after the intervention, and at 15 and 30 days post intervention.

Procedures Patients who meet the inclusion criteria will be invited to take part in the study by means of a study information sheet. Any doubts that may arise will be answered at the time.

Once informed, they will be asked to agree to be included in the study by signing the informed consent form, which will be given to them before starting the data collection.

After stratification of the patients, they will be randomised by balanced block randomisation into one of the following two groups:

Intervention group 1:

US-guided PNM with the conventional frequency of the Valera Minaya protocol, with localised location in the peripheral nerve. Stimulation of the superior gluteal nerve and inferior gluteal nerve will be performed, with 10 stimulations, with 10 seconds of stimulation and 10 seconds of rest, at a frequency of 10 Hz, with a pulse amplitude of 250 μs, and of maximum intensity tolerable by the patient that causes an exacerbated muscular contraction.

Intervention group 2:

High-frequency US-guided PNM with localised peripheral nerve location. Ten 10-second stimulations of the upper gluteal nerve and lower gluteal nerve will be performed, with frequency sweeps of 20Hz -100Hz with a pulse amplitude of 250 μs, and of maximum intensity tolerable by the patient that causes an exacerbated muscle contraction, with 10 seconds of rest between each stimulation.

US-guided PNM is a safe technique with minimal risk and is a technique used daily in clinical practice in physiotherapy clinics.

The procedure may cause temporary discomfort or slight prick pain during the act of puncture, which is performed with a very fine acupuncture needle.

Common adverse effects are local pain due to the puncture effect and small, short-lasting bruises.

Statistical analysis Baseline characteristics of the sample will be categorised, variables will be described as number, mean or median.

Comparison of demographic data and baseline measurements between the two groups will be compared using Student's t-test for independent samples or the Mann-Whithey U-test. Comparison of proportions shall be performed by applying binomial tests. The calculation of the degree of concordance between dichotomous variables by calculating the Kappa index.

The distribution of quantitative variables will be determined using the Kolmogrorov-Smirnov test. Analyses between and within intervention groups will be performed using a mixed model analysis of variance (ANOVA), for repeated measures with Bonferroni post hoc pairwise comparisons when a normal distribution is detected. Where a non-normal distribution is assumed, a non-parametric analysis will be performed, using the Mann-Whitney U-test for between-group comparisons and Tukey's test with Friedman's test to rule out within-group differences. An intention-to-treat analysis will be included to assess the possible dropout of subjects within the different groups.

Similarly, effect size will be calculated using Cohen's d o r to determine clinical significance: insignificant, small, medium and large differences will be reflected in effect sizes of <0.2 0.2-0.5 0.5-0.8 and >0.8, respectively.

The relationship between quantitative measures shall be determined by calculating Pearson's or Spearman's correlation coefficient as appropriate.

The confidence level of the statistical analysis shall be carried out at a 95% confidence level and a significant value shall be considered when p < 0.05. The statistical package SPSS for Windows, version 25 (SPSS, Chicago, IL) will be used.

Limitations of the study This study may be affected by the limitations of the responses of those undergoing treatment, appreciating that there are responders and non-responders when invasive techniques are applied.

There is blinding for the evaluator of the data, for the researcher conducting the assessment tests and for the patient him/herself. The degree of blinding obtained in the case of patients will be analysed.

The risk of measurement bias of all assessment tools, which will be mitigated by the use of ultrasound and the monitoring of the whole process in a carefully standardised way.

Subjects will participate freely and voluntarily without any coercion or pressure. The interventions performed during the assessment sessions do not involve any kind of rest except for possible discomfort related to the application of the puncture.

There are no published scientific studies that refer to the existence of risks and/or adverse effects with regard to the puncture intervention.

In reference to the puncture, studies have been published indicating its benefits without observing related risks. Nevertheless, adverse effects will be recorded if they occur.

Subjects will not receive any financial compensation for participation in the study and the authors of the project declare that they have no conflict of interest.

Data Protection legislation will be complied with at all times. Coded data will be used so that no subject data will be included in the study database and no one other than the research team will have access to the participant's identity. The collection and processing of data will be carried out electronically in accordance with the provisions of the General Data Protection Regulation (EU Regulation 2016/679) and Organic Law 3/2018, of 5 December, and participants are informed that the data provided will become part of a treatment for which the University of Zaragoza. Participants will be duly informed of all of the above and that they may at any time exercise their rights of access, rectification, suppression and portability of their data, as well as limitation and opposition to its processing, in accordance with the accompanying Information and Consent Document.

The researcher in charge of administering the interventions of the present project, through his membership of the College of Physiotherapists of Catalonia, has a civil liability policy that will be responsible for assuming liability in the event that the participants in the study suffer any damage or harm as a result of their participation. Policy number: 171676; Insurance company: RELYENS MUTUAL INSURANCE Sucursal en España, with C.I.F W0010878G and address at Paseo de la Castellana 110, Madrid 28046.

Adverse effects The US-guided PNM technique is an effective treatment procedure that is within the scope of physiotherapy practice. Education and training in physiotherapy provides practitioners with the anatomy, basic science and clinical basis to use this intervention safely and effectively. All invasive techniques have possible adverse effects that may arise from the intervention, which are typical of any intervention with puncture in the field of physiotherapy, and can be summarised as small bruises and short-lasting local pain due to the mechanical effect of the puncture.

No potential risks have been described so far, as these can be prevented by knowledge of the anatomy, training and experience of the operator. Significant adverse effects are rare. An overview of 17 systematic reviews of adverse events with consistent results shows that serious adverse effects may occur in as few as one in 100,000 needle insertions. Very rare and isolated cases of pneumothorax or serious infections have been reported.

Safe, evidence-based implementation of the procedure is based on a thorough understanding of the underlying anatomy and potential risks, and risks are coordinated with patients through informed consent.

Adverse effects arising from the intervention in this study will be monitored by the investigators and recorded within the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Healthy patients at the time of inclusion selection.
* Patients with a history of low back pain, without acute episodes at the time of the study.
* Patients who show an alteration in the function of the gluteus maximus and gluteus medius by EMG.
* Patients who show a decrease in the strength of the gluteus maximus and gluteus medius by dynamometry.
* Patients who have signed the information and consent document for participation.

Exclusion Criteria:

* Patients with belenophobia.
* Pregnant patients.
* Patients with cardiac pathologies or with pacemakers that do not allow electrical stimulation.
* Patients with low back pain in the acute phase.
* Patients with chronic low back pain.
* Patients with skin or immune disorders with contraindications for the application of invasive techniques.
* Patients who refuse to sign the informed consent or to participate in the study.
* Individuals who are planning a change in their lifestyle that involves a change in relation to physical activity or training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Dynamic strength gluteus | Baseline, immediately post intervention, 15 days post intervention, 30 days post intervention
  digital dynamometer, Wagner Force TenTM Digital Force Cage Algometer, FPX25, Massachusetts, USA.

SECONDARY OUTCOMES:
Isometric strenght gluteous | Baseline, immediately post intervention, 15 days post intervention, 30 days post intervention
  Isometric strenght gluteous, traction dynamometer (MicroFet2 hand-held dynamometer, Hoggan Health Industries, Biometrics, Netherlands) or (Force sensor, Chronojump, Boscosystem, Barcelona, Spain).
Contraction speed | Baseline, immediately post intervention, 15 days post intervention, 30 days post intervention
  Gluteus contraction speed (Encoder lineal Chronojump, Boscosystem, Barcelona, España).
Fatigue resistance | Baseline, immediately post intervention, 15 days post intervention, 30 days post intervention
  Gluteus fatigue resistance with repetitions
Power | Baseline, immediately post intervention, 15 days post intervention, 30 days post intervention
  Gluteus power (rotary encoder, Chronojump, Boscosystem, Barcelona, Spain)
Jump | Baseline, immediately post intervention, 15 days post intervention, 30 days post intervention
  Vertical jump parameters, with pressure platform (Contact platform, Chronojump, Boscosystem, Barcelona, Spain).
Reactivity | Baseline, immediately post intervention, 15 days post intervention, 30 days post intervention
  Reactivity in braking and exit time, with pressure platform (Contact platform, Chronojump, Boscosystem, Barcelona, Spain).
Range of motion | Baseline, immediately post intervention, 15 days post intervention, 30 days post intervention
  hip range motion with goniometer (Hawk-HCT digital goniometer, Human Computer Technology, Madrid, Spain).
Electromiography | Baseline, immediately post intervention, 15 days post intervention, 30 days post intervention
  Gluteus surface electromyography in isometric contraction and in dynamic contraction (mDurance System, mDurance Solutions, Granada, Spain)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Badia Rosells, Physiotherapist, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Fiostec Funcional, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-02-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT06873386/ICF_000.pdf